CLINICAL TRIAL: NCT00562224
Title: Phase I Dose-Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of PCI-24781 Administered Orally in Patients With Advanced Cancer
Brief Title: Study of the Safety and Tolerability of Oral Capsule Form of PCI-24781 in Advanced Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0402
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Neoplasms by Site; Lymphoma, Non-hodgkin; Hodgkin Disease; Multiple Myeloma; Leukemia, Lymphocytic, Chronic
Keywords: PCI-24781; Neoplasms by site; Lymphoma, non-hodgkin; Hodgkin disease; Multiple myeloma; Leukemia, lymphocytic, chronic
MeSH Terms: conditions — Neoplasms by Site; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — abexinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): All study subjects will receive PCI-24781 (study drug).
  Interventions: Drug: PCI-24781

INTERVENTIONS:
Drug: PCI-24781 — Up to 7 cohorts will receive PCI-24781 orally at doses starting at 30 mg/m2 three times a day approximately 4 hours apart ("TID"), up to 90 mg/m2, administered 5 days/week during the first 21 days of each 28 day cycle until MTD is reached. If a dose limiting toxicity (DLT) occurs, then the next cohort will receive PCI-24781 twice a day approximately 4 hours apart ("BID"). If a DLT occurs on the "BID" schedule, the subsequent cohort will receive PCI-24781 BID for 7 days every other week (2 times in a 28 day cycle). If a DLT occurs on this dosing schedule, then the next cohort will receive PCI-24781 BID for 5 days/week every other week (2 times in a 28 day cycle) until the maximum tolerated dose is reached.

SUMMARY:
To determine the highest dose of study drug that can be taken without causing serious side effects in patients with advanced cancer. The study will look at safety of the study drug and whether the treatment schedule is tolerated by patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Histologically confirmed, measurable solid tumor, non-Hodgkin's lymphoma, Hodgkin's disease, chronic lymphocytic leukemia, or multiple myeloma that has relapsed after standard therapy or for which no standard therapy exists
* Ability to swallow oral capsules without difficulty
* Estimated life expectancy > 12 weeks
* ECOG performance status ≤ 2
* Creatinine ≤ 1.5 × institutional upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 × institutional ULN (unless elevated from documented Gilbert's syndrome)
* AST and ALT ≤ 2.5 × institutional ULN (≤ 5 × institutional ULN in the presence of liver metastases)
* Platelet count ≥ 100,000/µL
* ANC ≥ 1500/µL
* Hgb ≥ 9.0 g/dL
* Patients with previously treated, stable, asymptomatic brain metastases who are not on corticosteroids are eligible
* Willing and able to sign a written informed consent-

Exclusion Criteria:

* Patients who have had immunotherapy, chemotherapy, or radiotherapy within 4 weeks (within 6 weeks for nitrosoureas or mitomycin C) prior to first day of drug dosing
* Patients who have undergone major surgery within 4 weeks prior to first day of drug dosing
* Patients who have received another investigational drug within 4 weeks
* Evidence of leptomeningeal metastasis
* Patients unable to swallow oral medications or with pre-existing gastrointestinal disorders that might interfere with proper absorption of the oral drugs (eg, WDHA syndrome, carcinoid syndromes, diarrhea due to infections, malabsorption syndromes secondary to surgery or chemotherapy)
* Uncontrolled illness including but not limited to: ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV heart failure), unstable angina pectoris, cardiac arrhythmia, and psychiatric illness that would limit compliance with study requirements
* Patients with risk factors for, or who are receiving medications known to prolong QTc interval and that may be associated with Torsades de Pointes
* QTc prolongation (defined as a QTc interval ≥ 450 msecs) or other significant ECG abnormalities including 2nd degree AV block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min).
* History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty and/or stenting within the past 6 months.
* Patients with known HIV infection
* Pregnant or lactating women (female patients of child-bearing potential must have a negative serum pregnancy test within 14 days of first day of drug dosing, or, if positive, a pregnancy ruled out by ultrasound)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity assessment at the end of the first 28 day cycle. | at the end of the first 28 day cycle

SECONDARY OUTCOMES:
Measure: Adverse event assessed through 30 days after last dose of study drug Measure: Tumor response Measure: Pharmacokinetic/Pharmacodynamic assessments | AE through 30 days after last dose of study drug, Tumor response at the end of every 2nd 28 day cycle, PK/PD assessments on Day 1, 2, 3 (or 4 or 5), and Day 8 of cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Samir Undevia, MD, Principal Investigator — University of Chicago
Locations (4):
- United States (4):
  - California Cancer Care, Greenbrae, California
  - University of Chicago, Chicago, Illinois
  - Sarah Cannon Research Institue, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Buggy JJ, Cao ZA, Bass KE, Verner E, Balasubramanian S, Liu L, Schultz BE, Young PR, Dalrymple SA. CRA-024781: a novel synthetic inhibitor of histone deacetylase enzymes with antitumor activity in vitro and in vivo. Mol Cancer Ther. 2006 May;5(5):1309-17. doi: 10.1158/1535-7163.MCT-05-0442. PMID 16731764
- See also: Related Info — http://www.pharmacyclics.com/